CLINICAL TRIAL: NCT00174135
Title: Sarcopenia Studies for the Elderly Population in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701210
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-08-30 (Estimated); Status verified 2004-12

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; exercise
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Health promotion in the elderly has been a major recent public health concern. Sarcopenia is a term utilized to define the loss of muscle mass and strength that occurs with aging. It has been demonstrated to be associated with decreased functional capacity among the elderly. The magnitude of the public health problem posed by sarcopenia is not yet established. The purposes of this study are to investigate sarcopenia and its relationship with functional status in elderly Taiwanese community-dwellers, and to develop the preventive strategy for sarcopenia in the elderly. Firstly, the investigators will recruit 100 volunteers (aged 18-90 years old) to participate in this study. All of the participants will receive bioelectric impedance analysis (BIA), muscle strength and endurance assessment, physical activity level assessment by a seven-day recall questionnaire, protein intake assessment, cognition evaluation (Mini-Mental State Examination) and functional status assessment by the Functional Independence Measurement (FIM) questionnaire. A multiple regression model will be used for statistical analyses. Then, this project will be used to evaluate the efficacy of a 12-week supervised resistance strengthening exercise program for sarcopenia in the elderly. Participants who are defined as having sarcopenia from the previous examination will be randomized into either the exercise or control groups. Subjects in the exercise group will receive resistance strengthening exercises 3 times per week for 12 weeks. All measurements will be performed as described above. The investigators expect that resistance exercises are effective in offsetting age-related decline of muscle mass and strength in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 year old healthy adults

Exclusion Criteria:

* No systemic diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Yueh Chien, MS, Principal Investigator — National Taiwan University, College of Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chien MY, Kuo HK, Wu YT. Sarcopenia, cardiopulmonary fitness, and physical disability in community-dwelling elderly people. Phys Ther. 2010 Sep;90(9):1277-87. doi: 10.2522/ptj.20090322. Epub 2010 Jul 8. PMID 20616117